CLINICAL TRIAL: NCT01520636
Title: What Should be the Best Physiotherapy Early After Stroke ?
Brief Title: Active MOBility Early After Stroke : What Should be the Best Physiotherapy Early After Stroke ?
Acronym: AMOBES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100124; 2011-A01049-32 (Other: IDRCB)
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2017-04

CONDITIONS: Rehabilitation
Keywords: stroke; early rehabilitation; motor recovery; functional recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1: standard physiotherapy (Placebo Comparator): daily physiotherapy aiming at preventing complications, going with the patient progress capacities, passive mobilisation, sitting as soon as possible, walking when possible, respiratory physiotherapy. 15-20 minutes total per day.
  Interventions: Procedure: standard physiotherapy
- group 2: experimental physiotherapy (Experimental): physiotherapy as described above added to verticalisation as soon as possible; active, intense and repeated motor exercises for limbs and trunk with all the available techniques. 60 minutes total per day.
  Interventions: Procedure: experimental physiotherapy

INTERVENTIONS:
Procedure: standard physiotherapy — daily physiotherapy aiming at preventing complications, going with the patient progress capacities, passive mobilisation, sitting as soon as possible, walking when possible, respiratory physiotherapy. 15-20 minutes total per day
  Arms: group 1: standard physiotherapy
Procedure: experimental physiotherapy — physiotherapy as described above added to verticalisation as soon as possible; active, intense and repeated motor exercises for limbs and trunk with all the available techniques. 60 minutes total per day.
  Arms: group 2: experimental physiotherapy

SUMMARY:
This study is designed to observe the respective effects of 2 types of physiotherapy early after a cerebral stroke. The hypothesis is that an intensive physiotherapy early delivered (Day 2 to D15) after a stroke could induce faster motor control recovery than a conservative physiotherapy aiming at preventing complications.

DETAILED DESCRIPTION:
Hypothesis:

An intensive and active physiotherapy delivered as soon as D2 post stroke could induce faster motor control recovery and autonomy than could do an usual conservative treatment aiming at preventing complications. The benefits could be a shortened inpatient stay (both in stroke unit and rehabilitation centre), a reduction of the secondary complications with a cut in of the total cost of care.

Primary objective:

To compare two strategies of physiotherapy on the evolution of motor control recovery during the first 3 months post stroke.

Secondary objectives :

To compare two strategies of physiotherapy on:

* Motor control deficiency on D15, D30, D45, M3
* Total length of stay as inpatient
* Autonomy on D15, D30, D45, M3
* Frequency of unexpected events
* Quality of life on M3
* Living place on M3

Assessment criteria:

-First criterion : Evolution of the motor control deficiency assessed by the Fugl Meyer (FM) scale modified by LINDMARK between day 0 and month 3.-Secondary criteria :

* Motor control deficiency assessed by the FM scale on D15, D30, D45, M3 and by the time requested before being able to walk 10 meters without human assistance.
* Total length of stay as inpatient
* Autonomy assessed by the Functional Independence Measure (motor subscale) on D30 and M3 and by the Rankin scale on D15, D30, D45, M3.
* Unexpected events recorded on D30 and M3
* Quality of life assessed by the Stroke Impact Scale on M3
* Residency

Method:

This is a "Zelen", single-blinded, randomised, controlled, multicentric trial aiming at comparing intensive physiotherapy after a stroke with the usually more conservative physiotherapy provided. Treatment is applied from the inclusion to the end of the stroke unit stay or until D15 post stroke.

* Group 1: daily physiotherapy aiming at preventing complications, going with the patient progress capacities, passive mobilisation, sitting as soon as possible, walking when possible, respiratory physiotherapy. 15-20 minutes total per day.
* Group 2: physiotherapy as described above added to verticalisation as soon as possible; active, intense and repeated motor exercises for limbs and trunk with all the available techniques. 60 minutes total per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients informed and giving their written consent.First
* Ever ischemic hemispheric or haemorrhagic stroke, unilateral, occurred between the 25th and the 72nd previous hours
* Age ≥ 18 years old
* Motricity quoted by an NIHSS >=2 in the upper limb or in the lower limb

Exclusion Criteria:

* Patient without health insurance.
* Coma (NIHSS consciousness > or = 2)
* Total recovery within the 24 first hours
* Brain stem or cerebellar stroke
* Previous neurological history, specially stroke or dementia
* Inability to understand the study
* Surgical treatment of the stroke
* Autonomy before stroke assessed by Rankin score different from 0
* Scheduled surgery in the following 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the motor control deficiency assessed by the Fugl Meyer (FM) scale modified by LINDMARK | between day 0 and month 3

SECONDARY OUTCOMES:
Motor control deficiency assessed by the FM scale | at D15, D30, D45, M3
  Motor control deficiency assessed by the FM scale on D15, D30, D45, M3 and by the time requested before being able to walk 10 meters without human assistance.
Total length of stay as inpatient | up to D30
  Total length of stay as inpatient
Autonomy assessed by the Functional Independence Measure (motor subscale) | at D30 and M3
Autonomy assessed by the Rankin scale | at D15, D30, D45, M3.
Unexpected events | at D30 and M3
  Unexpected events recorded on D30 and M3
Quality of life assessed by the Stroke Impact Scale | at M3
  Quality of life assessed by the Stroke Impact Scale on M3
Residency | at M3
Scale PASS | at D30 and M3
  Evaluation scale of balance PASS at D30 and M3

CONTACTS AND LOCATIONS:
Overall Officials: Alain YELNIK, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Service de MPR - Hôpital Fernand Widal, Paris
  - Service de Neurologie - Hôpital Lariboisière, Paris

REFERENCES:
- [Result] Yelnik AP, Quintaine V, Andriantsifanetra C, Wannepain M, Reiner P, Marnef H, Evrard M, Meseguer E, Devailly JP, Lozano M, Lamy C, Colle F, Vicaut E; AMOBES Group. AMOBES (Active Mobility Very Early After Stroke): A Randomized Controlled Trial. Stroke. 2017 Feb;48(2):400-405. doi: 10.1161/STROKEAHA.116.014803. Epub 2016 Dec 22. PMID 28008092